CLINICAL TRIAL: NCT01032538
Title: Time-dependent Improvement of Functional Outcome Following Oxford Medial Unicondylar Knee Replacement - A Prospective Longitudinal Study With Repetitive Measures of KOOS in 100 Patients
Brief Title: Time-dependent Improvement of Functional Outcome Following Oxford Medial Unicondylar Knee Replacement
Status: Completed | Type: Observational
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Tor Kjetil Nerhus, Consultant Orthopaedic surgeon, Vestre Viken Hospital Trust
Other Study IDs: TKN-002; 19441 (NSD) (Registry Identifier: Norwegian Privacy Ombudsman for Research)
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Osteoarthritis
Keywords: Unicondylar Knee Replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with knee osteoarthritis: Patients with knee osteoarthritis that are about to get an operation with oxford unicondylar knee

SUMMARY:
The objective of this prospective study is to determine (1) the time course of patient-relevant functional outcome evaluated by the Knee injury and Osteoarthritis Outcome Score (KOOS) and (2) the time course of range of motion (ROM) the first six years following Oxford Medial Unicondylar Knee prosthesis. Improvement of patient self-reported pain and daily function during the study period, are of particular interest.

DETAILED DESCRIPTION:
The objective of this prospective study is to determine (1) the time course of patient-relevant functional outcome evaluated by the Knee injury and Osteoarthritis Outcome Score (KOOS) and (2) the time course of range of motion (ROM) the first six years following Oxford Medial Unicondylar Knee prosthesis. Improvement of patient self-reported pain and daily function during the study period, are of particular interest. Thats it!

ELIGIBILITY:
Inclusion Criteria:

* patients with medial knee osteoarthritis
* admitted for unicondylar knee replacement
* age 50-80 years

Exclusion criteria

* rheumatoid arthritis
* previous knee infection

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients operated with total knee arthroplasty at Martina Hansens Hospital, Akershus University Hospital and Baerum hospital
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2003-11; Primary Completion 2009-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tor Kjetil Nerhus, MD, Principal Investigator — Martina Hansens Hospital
Locations (3):
- Norway (3):
  - Bærum Sykehus, Bærum, Akershus
  - Akershus University Hospital, Lørenskog, Akershus
  - Martina Hansens Hospital, Bærum, Bærum

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All recruited from Martina Hansens Hospitals patients
Groups:
- Patients With Knee Osteoarthritis: Patients eglible for unicondylar knee replacement
Period: Overall Study
Arm/Group | Patients With Knee Osteoarthritis
Started | 99 (Knees)
Completed | 99 (Knees)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Number of patients were 96. 3 patients were operated bilaterally. Number of knees were therefore 99.
Groups:
- Patients With Knee Osteoarthritis: Patients eglible for medial unicompartmental knee replacement
Arm/Group | Patients With Knee Osteoarthritis
Number analyzed (Participants) | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 39
Region of Enrollment [Number; unit: participants]
  Norway | 96

OUTCOME MEASURES:

1. Primary Outcome: Knee Injury and Osteoarthritis Outcome Score
Description: Patient relevant knee score. Validated score with 5 arms. 0-100, 100 is best.
Time Frame: Preoperative until 2 years postoperatively
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- KOOS Pain 2 Years: Knee pain score, one of 5 subscores of KOOS
- KOOS ADL 2 Years: Activities of dayly living score
Arm/Group | KOOS Pain 2 Years | KOOS ADL 2 Years
Number analyzed (Participants) | 96 | 96
units on a scale | 85.5 [82 to 89] | 88.2 [85 to 91]

2. Secondary Outcome: Range of Motion
Time Frame: Preoperative until 2 years postoperatively
Measure: Mean (95% Confidence Interval); unit: degrees
Groups:
- Passive ROM 2 Years: Range of motion measured by physiotherapist
Arm/Group | Passive ROM 2 Years
Number analyzed (Participants) | 96
degrees | 128 [123 to 130]

3. Secondary Outcome: Oxford Knee Score
Time Frame: Preoperative until 2 years postoperatively
Reporting Status: Not Posted

4. Secondary Outcome: UCLA Score
Time Frame: Preoperative until 2 years postoperatively
Reporting Status: Not Posted

5. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score
Time Frame: 10 years postoperatively
Reporting Status: Not Posted

6. Secondary Outcome: Oxford Knee Score
Time Frame: 10 years postoperatively
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: 96 patients with 99 knees included in the study
Groups:
- Patients With Knee Osteoarthritis: Patients eglible for unicompartmental knee replacement
Arm/Group | Patients With Knee Osteoarthritis
Serious Adverse Events (participants affected / at risk) | 5/96
Other Adverse Events (participants affected / at risk) | 0/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Knee Osteoarthritis (N=96)
Revision to total knee arthroplasty (Musculoskeletal and connective tissue disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No